CLINICAL TRIAL: NCT03184831
Title: Comparison of Deproteinized Bovine Bone Mixed With Injectable Platelet Rich Fibrin Versus a Sole Deproteinized Bovine Bone "TUTOGEN BONE" in Sinus Floor Elevation With Simultaneous Implant Placement. A Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ali El Sayed Attia, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cebc.CairoUniver
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Sinus Floor Elevation
Keywords: sinus lift, injectable platelet rich fibrin, sticky bone, bovine bone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sinus lift, implant placement, sole bovine bone (Active Comparator): sinus floor elevation with simultaneous implant placement together with grafting the sinus with a deproteinized bovine bone solely.
  Interventions: Procedure: sinus lift, implant placement, sole bovine bone
- sinus lift, implant placement, injectable PRF + bovine bone (Experimental): sinus floor elevation with simultaneous implant placement together with grafting the sinus with a mixture of injectable platelet rich fibrin with a deproteinized bovine bone.
  Interventions: Procedure: sinus lift, implant placement, injectable PRF + bovine bone

INTERVENTIONS:
Procedure: sinus lift, implant placement, sole bovine bone — sinus lift augmentation with a sole deproteinized bovine bone with simultaneous implant placement
  Arms: sinus lift, implant placement, sole bovine bone
Procedure: sinus lift, implant placement, injectable PRF + bovine bone — sinus lift augmentation with a mixture of injectable platelet rich fibrin plus a deproteinized bovine bone with simultaneous implant placement
  Arms: sinus lift, implant placement, injectable PRF + bovine bone

SUMMARY:
28 recruited patients indicated for sinus floor elevation with simultaneous implant placement . they were divided into two groups. first group was assigned for placement of deproteinized bovine bone solely, while the other group was assigned for the placement of mixture of injectable platelet rich fibrin with deproteinized bovine bone into the sinus after implant placement.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring implants in maxilla and have atrophic bone regarding the length due to sinus pneumatiztion. Length 3: 7 mm .

Exclusion Criteria:

1. General contraindications for implant
2. Systemic diseases that might affect the healing of bone
3. Patients with sinus pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 7 days postoperative
  evaluation of postoperative complications in terms of pain and edema using patient pain chart

SECONDARY OUTCOMES:
implant stability | will be measured intraoperatively immediately after insertion of the implant and will be measured one more time 6 months after the first operation at time of implant exposure
  measurement of implant stability using osstell device
height of bone gained around the implant | 6 months postoperative
  two cone beam computed tomography (CBCT) will be taken one immediate postoperative and the other 6 months after the first operation then the height of bone gained around the implant will be assessed by superimposing the same sections in the two CBCT
bone density around the implant | 6 months postoperative
  Bone density will be measured by calculating the difference in the Hounsfield unit (HU) in the bone around the implants in the immediate postoperative CBCT (within one week) and the CBCT after 6 months.

IPD SHARING:
Plan to Share IPD: Undecided